CLINICAL TRIAL: NCT01424410
Title: Health Benefits of Repeated Treatment in Pediatric Schistosomiasis
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); University of Zimbabwe (Other)
Responsible Party: Principal Investigator, Dr Francisca Mutapi, Dr, University of Edinburgh
Other Study IDs: ERI019729-THRASHER
Record Dates: First submitted 2011-06-16; First posted 2011-08-29 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Schistosomiasis
Keywords: paediatric schistosomiasis morbidity immunology
MeSH Terms: conditions — Schistosomiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Objective and Hypotheses: This project has the overall objective of implementing and evaluating new approaches to reducing the current and future burden of urinary schistosomiasis in young children using the antihelminthic drug praziquantel. The investigators hypotheses are that (1) praziquantel treatment will be as effective in children 1 to 5 years of age (who are routinely excluded from schistosomiasis control programmes) as it is in older 6-10 year old children and (2) two treatments will be more effective than a single treatment, especially in children 1 to 5 years of age.

DETAILED DESCRIPTION:
This study aims to address the present health inequity by refinement of an existing drug regimen to improve the current and future health of pre-school children and infants. Praziquantel is cheap, highly efficacious and safe, presenting a realistic opportunity of using a pre-existing tool in a modified way to benefit child health and development. The study will focus on children aged 1 to 10 years of age, comparing the impact of single vs. double treatment with PZQ on the current and future health status of the children. The immediate health benefits of PZQ treatment in children aged 6-10 years of age have already been documented and therefore by including 6-10 year olds in the proposed study, we can determine if the effects of PZQ treatment on health and morbidity measures is age dependent. By killing worms PZQ stops the morbidity related to the presence of worms and eggs such as anaemia, abdominal pain, diarrhoea and blood in the urine. Therefore the study will investigate the immediate health benefits of treating pre-school children and infants.

ELIGIBILITY:
Inclusion Criteria:

1. lifelong residents of the area
2. have provided at least 2 urine and 2 stool for parasitological examination
3. have given a blood sample before and after each treatment episode
4. be negative for hookworm, Trichuris and Ascaris

Exclusion Criteria:

1. clinical signs of tuberculosis or malaria
2. presenting with fever
3. have had a recent major operation, illness or vaccination
4. have previously received antihelminthic treatment

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Zimbabwean children
Sampling Method: Non-Probability Sample
Enrollment: 360 (Actual)
Dates: Start 2012-02; Primary Completion 2014-07 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in schistosome-specific and systemic immune responses | 6 weeks
  Determine the change at 6 weeks post antihelminthic treatment from baseline of schistosome-specific and systemic immune responses

SECONDARY OUTCOMES:
Change from baseline in schistosome-specific and systemic immune responses | 12 months
  Determine the change at 12 months post antihelminthic treatment from baseline of schistosome-specific and systemic immune responses. Determine the effects of single and double antihelminthic treatments on these immunological changes.
Change from baseline in schistosome-related morbidity and disease markers | 6 weeks
  Determine the change in prevalance and magnitude of schistosome-related disease and morbidity markers at 6 weeks from those at baseline.
Change from baseline in morbidity and disease markers | 12 months
  Determine the change in prevalance and magnitude of schistosome-related disease and morbidity markers at 12 months from those at baseline. Determine the effects of single and double antihelminthic treatments on the disease and morbidity measures.

CONTACTS AND LOCATIONS:
Overall Officials: Francisca Mutapi, PhD, Principal Investigator — University of Edinburgh
Locations (1):
- National Institutes for Health Research, Harare, Zimbabwe

REFERENCES:
- [Background] Wami WM, Nausch N, Bauer K, Midzi N, Gwisai R, Simmonds P, Mduluza T, Woolhouse M, Mutapi F. Comparing parasitological vs serological determination of Schistosoma haematobium infection prevalence in preschool and primary school-aged children: implications for control programmes. Parasitology. 2014 Dec;141(14):1962-70. doi: 10.1017/S0031182014000213. Epub 2014 Mar 28. PMID 24679476
- [Background] Mduluza T, Mutapi F. Putting the treatment of paediatric schistosomiasis into context. Infect Dis Poverty. 2017 Apr 7;6(1):85. doi: 10.1186/s40249-017-0300-8. PMID 28388940
- [Result] Wami WM, Nausch N, Midzi N, Gwisai R, Mduluza T, Woolhouse M, Mutapi F. Identifying and evaluating field indicators of urogenital schistosomiasis-related morbidity in preschool-aged children. PLoS Negl Trop Dis. 2015 Mar 20;9(3):e0003649. doi: 10.1371/journal.pntd.0003649. eCollection 2015 Mar. PMID 25793584
- See also: PI's webpage — http://pig.bio.ed.ac.uk/